CLINICAL TRIAL: NCT06860763
Title: Clinical Study on Acupuncture Treatment for Attention Deficit Hyperactivity Disorder.
Brief Title: Acupuncture for ADHD: Acupoint Data Mining, Clinical Effectiveness, and Interviews to Explore Treatment Outcomes.
Acronym: ACU-ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated Hospital of Beijing University of Chinese Medicine (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Principal Investigator, Tananan Sangwanit, Principal Investigator (PI), The Third Affiliated Hospital of Beijing University of Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BZYSY-2024YJSKTPJ-99
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-06

CONDITIONS: Acupuncture; ADHD - Attention Deficit Disorder With Hyperactivity; Children; Interview; Executive Functioning; Quality of Life (QOL)
Keywords: Acupuncture; ADHD; Executive functioning; Interview; TCM; PedsQL
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese Herbal Medicine (Active Comparator): Chinese herbal decoction based on the 2019 edition of the "Clinical Diagnosis and Treatment Guidelines for Pediatric ADHD" by the Chinese Society of Traditional Chinese Medicine.
  Interventions: Drug: Chinese herbal medicine
- Acupuncture (Experimental): Acupuncture will be based on the first phase of data analysis, which identifies acupuncture point selection patterns for ADHD in school-age children.
  Interventions: Drug: Chinese herbal medicine; Device: Acupuncture

INTERVENTIONS:
Drug: Chinese herbal medicine — The general treatment strategy will follow principles of clearing excess and replenishing deficiency, regulating the internal organs, and balancing yin and yang. Based on the patient's specific syndrome in TCM.
Device: Acupuncture — The acupuncture needles used will be 0.25 mm in diameter and 25 mm in length, inserted quickly with even supplementation and reduction techniques.
  Arms: Acupuncture

SUMMARY:
This study aims to evaluate the efficacy of acupuncture as a treatment for Attention Deficit Hyperactivity Disorder (ADHD) in children aged 6-12 years. Using a mixed-methods approach, the research will triangulate data from acupoint data mining, treatment outcomes assessment, and patient perspectives to provide a comprehensive analysis of acupuncture's potential therapeutic benefits for ADHD.

This prospective cohort study will recruit children diagnosed with ADHD, assigning them to receive either acupuncture combined with traditional Chinese herbal treatment or herbal treatment alone. Quantitative assessments using the the SNAP-IV, Conners 3-P, BRIEF-2, PedsQL™ 4.0 Generic Core Scales, PSQI and CGI that will be complemented by qualitative interviews to capture nuanced patient experiences and treatment outcomes.

The study will span 12 months, commencing on March 1st, 2025 with an expected completion by February 28th, 2026. By integrating quantitative assessments with qualitative insights, it aims to provide comprehensive evidence on acupuncture's role in ADHD management. Findings may inform clinical guidelines and enhance patient-centered care approaches.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) remains a prevalent neurodevelopmental disorder affecting children worldwide, often characterized by persistent patterns of inattention, hyperactivity, and impulsivity that significantly impair daily functioning. While conventional treatments such as stimulant medications and behavioral therapies are commonly prescribed, interest in complementary and alternative approaches, including acupuncture, has grown. This study proposes a rigorous examination of acupuncture's potential efficacy as a treatment modality for ADHD, employing a mixed-methods approach to triangulate acupoint data mining, treatment outcomes assessment, and patient perspectives.

The primary objective is to evaluate the therapeutic effects of acupuncture in children aged 6-12 years diagnosed with ADHD. The research design involves a prospective cohort study wherein participants will be allocated to receive either acupuncture combined with traditional Chinese herbal treatment or herbal treatment alone. Quantitative assessment of ADHD symptom and related impairment administered at baseline, post-treatment, and follow-up intervals. Additionally, qualitative interviews with participants, their caregivers and clinicians will explore subjective experiences, treatment satisfaction, and perceived changes in ADHD symptoms.

This prospective cohort study will recruit 6-12 year-old children diagnosed with ADHD from pediatrics department of the third affiliated hospital of Beijing University of Chinese Medicine. Participants will be randomly assigned to two groups: an experimental group receiving acupuncture alongside traditional Chinese herbal treatment, and a control group receiving only the herbal treatment. The study will adhere to ethical guidelines, ensuring informed consent from parents and assent from children.

The research content includes three parts, as follows Phase I: Acupoint data mining for core acupoints Acupoint data mining will guide personalized treatment protocols, selecting points historically used for ADHD and supported by current research.

Phase II: Clinical Trial Intervention Quantitative assessment will involve administering the SNAP-IV, Conners 3-P, BRIEF-2, PedsQL™ 4.0 Generic Core Scales, PSQI and CGI at baseline, post-treatment, and follow-up intervals to measure changes in ADHD symptomatology, executive function, quality of life, and sleep quality.

Phase III: Qualitative Interview Qualitative methods will complement quantitative findings, capturing subjective experiences through semi-structured interviews with children, parents, and clinicians. This approach aims to provide a holistic understanding of treatment efficacy, patient satisfaction, and perceived improvements in ADHD symptoms, executive function, quality of life, and sleep patterns.

Statistical analyses will compare SNAP-IV, Conners 3-P, BRIEF-2, PSQI and PedsQL™ 4.0 Generic Core Scales scores between groups, supplemented by thematic analysis of qualitative data to explore treatment satisfaction and symptom changes.

Statistical analyses, including paired t-tests, ANOVA, and thematic analysis, will be employed to compare outcomes between treatment groups and explore correlations between acupuncture treatment, symptom alleviation, and overall well-being measures.

ELIGIBILITY:
Inclusion Criteria:

Patients will be considered for enrolment if they meet the criteria of:

* A confirmed diagnosis of ADHD based on the DSM-5 criteria for ADHD (Western medical diagnosis) and in accordance with the ADHD Chinese Medicine Clinical Trial Design and Evaluation Technical Guidelines.
* Aged between 6 and 12 years.
* No use of any other pharmacological treatments (both Western and traditional Chinese medicine) within the two weeks prior to the start of the study.
* An IQ score of greater than 80, as determined by the Raven's Progressive Matrices test.
* The participant has not participated in any other clinical trials.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

* Do not meet the inclusion criteria
* Have comorbid psychiatric disorders, severe medical or psychiatric conditions that may interfere with the study (e.g., epilepsy, severe anxiety), pervasive developmental disorders, intellectual disability, or a history of suicidal or self-harming behavior
* Have participated in any other drug clinical trials within the past 3 months.
* Have severe comorbid conditions such as cardiovascular, hepatic, renal, or hematologic diseases.
* Have any other conditions that the researchers believe may interfere with the assessment of treatment efficacy or safety.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
SNAP-IV | From enrollment to the end of treatment at 8 weeks
  Swanson, Nolan, and Pelham Rating Scale.
  * Items: 18 (9 inattention + 9 hyperactivity/impulsivity).
  * Response Options: 0 = Not at all, 1 = Just a little, 2 = Quite a bit, 3 = Very much.
  * Interpretation: Higher scores mean more severe ADHD symptoms (worse outcome).

SECONDARY OUTCOMES:
Conners 3-P | From enrollment to the end of treatment at 8 weeks
  Conners 3rd Edition-Parent Rating Scale.
  * Items: 48
  * Response Options: 0 (Not true at all) to 3 (Very much true)
  * Interpretation: Higher scores reflect more severe ADHD-related problems (worse outcome)
BRIEF-2 | From enrollment to the end of treatment at 8 weeks
  Behavior Rating Inventory of Executive Function, Second Edition.
  * Items: 63
  * Response Options: 0 (Never) to 2 (Always)
  * Scoring: Raw scores are converted to T-scores; T-scores over 65 indicate a clinically elevated level
  * Interpretation: Higher T-scores denote greater executive function difficulties (worse outcome)
PedsQL 4.0 generic score | From enrollment to the end of treatment at 8 weeks
  Pediatric Quality of Life Inventory.
  * Items: 23
  * Response Options: 0 (Never), 2 (Sometimes), 4 (Always). Score Range: Original responses are transformed into a 0-100 scale
  * Interpretation: Higher scores indicate better quality of life (better outcome)
PSQI | From enrollment to the end of treatment at 8 weeks
  Pittsburgh Sleep Quality Index.
  * Items: 18 total
  * Response Options: For 14 of those items, 0 (Never), 1 (<1 time/week), 2 (2 times/week), 3 (≥3 times/week)
  * Score Range: 0-21 for the global score
  * Interpretation: Higher scores indicate poorer sleep quality (worse outcome)
VADRS | From enrollment to the end of treatment at 8 weeks
  Vanderbilt ADHD Diagnostic Rating Scale.
  * Items: 55 (ADHD core symptoms + comorbid items)
  * Response Options: 0 (Never) to 3 (Very often)
  * Interpretation: Higher scores signify more severe ADHD symptoms and comorbidity (worse outcome)
CGI | From enrollment to the end of treatment at 8 weeks
  Clinical Global Impression.
  CGI-Severity (CGI-S):
  * Scale: 7 points, typically from 1 (Normal, not ill) to 7 (Among the most extremely ill)
  * Interpretation: Higher scores indicate more severe illness (worse outcome).
  CGI-Improvement (CGI-I):
  * Scale: 7 points, typically from 1 (Very much improved) to 7 (Very much worse)
  * Interpretation: Lower scores indicate greater improvement, while higher scores represent worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Cui, Ph.D.,Prof., Study Director — Third Hospital of Beijing University of Chinese Medicine
Locations (1):
- Pediatrics Outpatient Department of the Third Affiliated Hospital of Beijing University of Chinese Medicine, Beijing, Chaoyang District, China

IPD SHARING:
Plan to Share IPD: No
Sharing IPD is not permitted due to privacy concerns, ethical and legal restrictions, and institutional policies. Protecting minors' confidentiality and adhering to data security standards are priorities.

REFERENCES:
- [Background] Casebeer AL, Verhoef MJ. Combining qualitative and quantitative research methods: considering the possibilities for enhancing the study of chronic diseases. Chronic Dis Can. 1997;18(3):130-5. PMID 9375260
- [Background] Zhao FY, Fu QQ, Kennedy GA, Conduit R, Zhang WJ, Wu WZ, Zheng Z. Can acupuncture improve objective sleep indices in patients with primary insomnia? A systematic review and meta-analysis. Sleep Med. 2021 Apr;80:244-259. doi: 10.1016/j.sleep.2021.01.053. Epub 2021 Feb 2. PMID 33610071
- [Background] Li S, Yu B, Lin Z, Jiang S, He J, Kang L, Li W, Chen X, Wang X. Randomized-controlled study of treating attention deficit hyperactivity disorder of preschool children with combined electro-acupuncture and behavior therapy. Complement Ther Med. 2010 Oct;18(5):175-83. doi: 10.1016/j.ctim.2010.08.002. Epub 2010 Aug 30. PMID 21056840
- [Background] Zhang L, Huang C, Chen X, Du S, Yang J, Hu B. The efficacy of acupuncture for attention deficit hyperactivity disorder (ADHD): An overview of systematic reviews and meta-analyses. Complement Ther Med. 2023 Sep;76:102968. doi: 10.1016/j.ctim.2023.102968. Epub 2023 Aug 8. PMID 37562658
- [Background] Ang L, Kim JT, Kim K, Lee HW, Choi JY, Kim E, Lee MS. Acupuncture for Treating Attention Deficit Hyperactivity Disorder in Children: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2023 Feb 17;59(2):392. doi: 10.3390/medicina59020392. PMID 36837594
- [Background] Zhou W, Cheng X, Zhang Y. Effect of Liuwei Dihuang decoction, a traditional Chinese medicinal prescription, on the neuroendocrine immunomodulation network. Pharmacol Ther. 2016 Jun;162:170-8. doi: 10.1016/j.pharmthera.2016.02.004. Epub 2016 Feb 16. PMID 26896567
- [Background] Wolraich ML, Hagan JF, Allan C, et al; Subcommittee on Children and Adolescents with Attention-Deficit/Hyperactive Disorder. Clinical Practice Guideline for the Diagnosis, Evaluation, and Treatment of Attention-Deficit/Hyperactivity Disorder in Children and Adolescents. Pediatrics. 2019;144(4):e20192528. Pediatrics. 2020 Mar;145(3):e20193997. doi: 10.1542/peds.2019-3997. No abstract available. PMID 32111626
- [Background] Langberg JM, Molitor SJ, Oddo LE, Eadeh HM, Dvorsky MR, Becker SP. Prevalence, Patterns, and Predictors of Sleep Problems and Daytime Sleepiness in Young Adolescents With ADHD. J Atten Disord. 2020 Feb;24(4):509-523. doi: 10.1177/1087054717690810. Epub 2017 Feb 4. PMID 28162039
- [Background] Liang X, Qiu H, Li SX. Objectively measured sleep continuity in children and adolescents with ADHD: A systematic review and meta-analysis. Psychiatry Res. 2023 Oct;328:115447. doi: 10.1016/j.psychres.2023.115447. Epub 2023 Aug 28. PMID 37657199
- [Background] Wanni Arachchige Dona S, Badloe N, Sciberras E, Gold L, Coghill D, Le HND. The Impact of Childhood Attention-Deficit/Hyperactivity Disorder (ADHD) on Children's Health-Related Quality of Life: A Systematic Review and Meta-Analysis. J Atten Disord. 2023 Apr;27(6):598-611. doi: 10.1177/10870547231155438. Epub 2023 Feb 17. PMID 36800919
- [Background] Danckaerts M, Sonuga-Barke EJ, Banaschewski T, Buitelaar J, Dopfner M, Hollis C, Santosh P, Rothenberger A, Sergeant J, Steinhausen HC, Taylor E, Zuddas A, Coghill D. The quality of life of children with attention deficit/hyperactivity disorder: a systematic review. Eur Child Adolesc Psychiatry. 2010 Feb;19(2):83-105. doi: 10.1007/s00787-009-0046-3. Epub 2009 Jul 26. PMID 19633992
- [Background] Groves NB, Wells EL, Soto EF, Marsh CL, Jaisle EM, Harvey TK, Kofler MJ. Executive Functioning and Emotion Regulation in Children with and without ADHD. Res Child Adolesc Psychopathol. 2022 Jun;50(6):721-735. doi: 10.1007/s10802-021-00883-0. Epub 2021 Nov 11. PMID 34762251
- [Background] Kofler MJ, Irwin LN, Soto EF, Groves NB, Harmon SL, Sarver DE. Executive Functioning Heterogeneity in Pediatric ADHD. J Abnorm Child Psychol. 2019 Feb;47(2):273-286. doi: 10.1007/s10802-018-0438-2. PMID 29705926
- [Background] Choi WS, Woo YS, Wang SM, Lim HK, Bahk WM. The prevalence of psychiatric comorbidities in adult ADHD compared with non-ADHD populations: A systematic literature review. PLoS One. 2022 Nov 4;17(11):e0277175. doi: 10.1371/journal.pone.0277175. eCollection 2022. PMID 36331985
- [Background] Anastopoulos AD, DuPaul GJ, Weyandt LL, Morrissey-Kane E, Sommer JL, Rhoads LH, Murphy KR, Gormley MJ, Gudmundsdottir BG. Rates and Patterns of Comorbidity Among First-Year College Students With ADHD. J Clin Child Adolesc Psychol. 2018 Mar-Apr;47(2):236-247. doi: 10.1080/15374416.2015.1105137. Epub 2016 Feb 6. PMID 26852645
- [Background] Danielson ML, Bitsko RH, Ghandour RM, Holbrook JR, Kogan MD, Blumberg SJ. Prevalence of Parent-Reported ADHD Diagnosis and Associated Treatment Among U.S. Children and Adolescents, 2016. J Clin Child Adolesc Psychol. 2018 Mar-Apr;47(2):199-212. doi: 10.1080/15374416.2017.1417860. Epub 2018 Jan 24. PMID 29363986
- [Background] Li F, Cui Y, Li Y, Guo L, Ke X, Liu J, Luo X, Zheng Y, Leckman JF. Prevalence of mental disorders in school children and adolescents in China: diagnostic data from detailed clinical assessments of 17,524 individuals. J Child Psychol Psychiatry. 2022 Jan;63(1):34-46. doi: 10.1111/jcpp.13445. Epub 2021 May 21. PMID 34019305
- [Background] Simon V, Czobor P, Balint S, Meszaros A, Bitter I. Prevalence and correlates of adult attention-deficit hyperactivity disorder: meta-analysis. Br J Psychiatry. 2009 Mar;194(3):204-11. doi: 10.1192/bjp.bp.107.048827. PMID 19252145
- [Background] Gao Q, Qian Y, He XX, Sun L, Chang WL, Li YL, Cao QJ, Wang YF, Qian QJ. Childhood predictors of persistent ADHD in early adulthood: Results from the first follow-up study in China. Psychiatry Res. 2015 Dec 30;230(3):905-12. doi: 10.1016/j.psychres.2015.11.025. Epub 2015 Nov 17. PMID 26614011